CLINICAL TRIAL: NCT01297985
Title: Efficacy of Peer-Led Education in Improving Mental Health Recovery Outcomes in Tennessee
Brief Title: A Randomized Controlled Trial of Mental Health Peer-Led Education
Acronym: BRIDGES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Judith A. Cook, Professor of Psychiatry, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2006-0024; H133B050003b (Other Grant/Funding Number: Nat'l Inst on Disability & Rehab Research, US Dept of Educ)
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Mental Disorders
Keywords: Serious mental illness; Psychiatric disability; Mental health peer-led; Mental illness education; Illness self-management
MeSH Terms: conditions — Mental Disorders | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BRIDGES Intervention (Experimental): The BRIDGES program is a 10-week, manualized education course designed to provide basic education about the etiology and treatment of mental illness, self-help skills, and recovery principles in order to empower participants to return to valued social roles within their communities. BRIDGES is a peer-led program and all instructors are adults with mental illnesses. For this intervention study, the BRIDGES curriculum was modified from a 10-week course to an 8-week course, meeting for 2 1/2 hours once a week.
  Interventions: Behavioral: BRIDGES Peer-Led Education
- Comparison Wait-list Group (No Intervention): Participants assigned to the comparison group were in a delayed treatment condition in which they continued in public services as usual, but were offered the chance to attend the BRIDGES program after their final research interview.

INTERVENTIONS:
Behavioral: BRIDGES Peer-Led Education — The BRIDGES program is a 10-week, manualized education course designed to provide basic education about the etiology and treatment of mental illness, self-help skills, and recovery principles in order to empower participants to return to valued social roles within their communities. BRIDGES is a peer-led program and all instructors are adults with mental illnesses. For this intervention study, the BRIDGES curriculum was modified from a week course to an 8-week course, meeting for 2 1/2 hours once a week.
  Other Names: Building Recovery of Individual Dreams and Goals through Education and Support
  Arms: BRIDGES Intervention

SUMMARY:
This randomized controlled trial tests the efficacy of a mental health peer-led educational intervention called BRIDGES (Building Recovery of Individual Dreams and Goals through Education and Support). The BRIDGES program is a 10-week, manualized education course designed to provide basic information about the etiology and treatment of mental illness, self-help skills, and recovery principles in order to empower participants to return to valued social roles within their communities. BRIDGES is a peer-led program and all instructors are adults with mental illnesses. For study purposes, the 10-week course was modified to 8-weeks, meeting 2 1/2 hours once a week.

Hypothesis #1: Compared to wait-list controls, intervention participants will report increased feelings of psychological empowerment.

Hypothesis #2: Compared to wait-list controls, intervention participants will report increased feelings of hopefulness.

Hypothesis #3: Compared to wait-list controls, intervention participants will report enhanced coping ability.

Hypothesis #4: Compared to wait-list controls, intervention participants will report enhanced recovery.

Hypothesis #5: Compared to wait-list controls, intervention participants will report greater ability to advocate for themselves with health care providers.

Hypothesis #6: Compared to wait-list controls, those in the BRIDGES education course will report increased knowledge of the causes and treatment of mental illness and recovery principles.

DETAILED DESCRIPTION:
Eligibility criteria included having a diagnosis of serious mental illness and experiencing severe functional impairment in one or more life roles. All study participants completed telephone interviews at three points in time: study entry (pre-intervention); 8-weeks later (immediate post-intervention); and 6-months after intervention (approximately 8 months after study entry). Blinded interviewers administered valid and reliable outcome assessments that measured changes in subjects' knowledge about mental illness; emotional well-being; empowerment; hopefulness; self-advocacy; and recovery. All study participants were compensated for their time at each interview. All BRIDGES instructors were people in recovery from serious mental illnesses who were certified and experienced BRIDGES teachers. Fidelity to the BRIDGES curriculum was assessed on an ongoing basis throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mental illness
* Disability due to mental illness
* Age 18 years or older
* Willingness to receive the intervention

Exclusion Criteria:

* Inability to understand spoken English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2006-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Cook, PhD, Principal Investigator — Department of Psychiatry, University of Illinois at Chicago; Susan A Pickett, PhD, Study Director — Department of Psychiatry, University of Illinois at Chicago
Locations (1):
- National Alliance on Mental Illness Tennessee, Nashville, Tennessee, United States

REFERENCES:
- [Background] Pickett SA, Diehl S, Steigman PJ, Prater JD, Fox A, Cook JA. Early outcomes and lessons learned from a study of the Building Recovery of Individual Dreams and Goals through Education and Support (BRIDGES) program in Tennessee. Psychiatr Rehabil J. 2010 Autumn;34(2):96-103. doi: 10.2975/34.2.2010.96.103. PMID 20952362
- [Result] Pickett SA, Diehl SM, Steigman PJ, Prater JD, Fox A, Shipley P, Grey DD, Cook JA. Consumer empowerment and self-advocacy outcomes in a randomized study of peer-led education. Community Ment Health J. 2012 Aug;48(4):420-30. doi: 10.1007/s10597-012-9507-0. Epub 2012 Mar 30. PMID 22460927
- [Result] Cook JA, Steigman P, Pickett S, Diehl S, Fox A, Shipley P, MacFarlane R, Grey DD, Burke-Miller JK. Randomized controlled trial of peer-led recovery education using Building Recovery of Individual Dreams and Goals through Education and Support (BRIDGES). Schizophr Res. 2012 Apr;136(1-3):36-42. doi: 10.1016/j.schres.2011.10.016. Epub 2011 Nov 29. PMID 22130108
- [Result] Steigman PJ, Pickett SA, Diehl SM, Fox A, Grey DD, Shipley P, Cook JA. Psychiatric symptoms moderate the effects of mental illness self-management in a randomized controlled trial. J Nerv Ment Dis. 2014 Mar;202(3):193-9. doi: 10.1097/NMD.0000000000000098. PMID 24566504

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted collaboratively with the statewide consumer coalition, Tennessee Mental Health Consumer's Association (TMHCA), and the statewide National Alliance for Mental Illness (NAMI), NAMI Tennessee. Recruitment took place from March 2007 through March 2009 at local mental health agencies, and at residential and peer-run programs.
Groups:
- BRIDGES Intervention: BRIDGES Peer-Led Education: The BRIDGES program is a 10-week, manualized education course designed to provide basic education about the etiology and treatment of mental illness, self-help skills, and recovery principles in order to empower participants to return to valued social roles within their communities. BRIDGES is a peer-led program and all instructors are adults with mental illnesses. For this intervention study, the BRIDGES curriculum was modified from a 10-week course to an 8-week course, meeting for 2 1/2 hours once a week.
Period: Overall Study
Arm/Group | BRIDGES Intervention | Comparison Wait-list Group
Started | 212 | 216
Completed | 157 | 163
Not Completed | 55 | 53

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BRIDGES Intervention | Comparison Wait-list Group | Total
Number analyzed (Participants) | 212 | 216 | 428
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.7 (9.9) | 43.0 (11.8) | 42.8 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 124 | 238
  Male | 98 | 92 | 190
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 75 | 71 | 146
  Not Hispanic or Latino | 137 | 145 | 282
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 15 | 25
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 75 | 71 | 146
  White | 112 | 117 | 229
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 11 | 9 | 20
Region of Enrollment [Number; unit: participants]
  United States | 212 | 216 | 428

OUTCOME MEASURES:

1. Primary Outcome: Recovery From Mental Illness
Description: Recovery from mental illness is measured by the Recovery Assessment Scale (RAS) (Giffort et al., 1995). Recovery is a psychosocial outcome assessed via patient self-ratings on a 41-item scale using a 5-point Likert-response format ranging from "strongly disagree" to "strongly agree." The minimum value for the RAS is 41 and the maximum is 205, with higher scores indicating a better outcome. Dimensions of recovery include personal confidence and hope, willingness to ask for help, goal and success orientation, reliance on others, and no being dominated by one's residual psychiatric symptoms.
Time Frame: Study entry (Pre-intervention/T1), 8-weeks later (Post-Intervention 1/T2), & 6-months after T2 (Post-Intervention 2/T3)
Population: The "Overall Number of Participants Analyzed" reflects the number of participants at Time 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BRIDGES Intervention | Comparison Wait-list Group
Number analyzed (Participants) | 212 | 216
score on a scale
  Baseline | 91.90 (13.65) | 90.72 (13.33)
  Post-intervention 1 (Time 2): number analyzed (Participants) | 170 | 171
  Post-intervention 1 (Time 2) | 94.84 (12.83) | 91.01 (14.35)
  Post-intervention 2 (Time 3): number analyzed (Participants) | 157 | 159
  Post-intervention 2 (Time 3) | 96.13 (12.76) | 91.97 (14.58)
Statistical Analysis 1: Comparison: BRIDGES Intervention vs Comparison Wait-list Group; This mixed effects random regression analysis tested whether intervention participants would report larger increases than controls in self-perceived Recovery and that this effect would be maintained overtime; and that intervention participants would report greater increases in hopefulness than controls, also maintained longitudinally This first model reports on Recovery over time; Test type: Superiority; p = .013, Mixed Effects Random Regression; MIXREG Estimate = 1.55, Standard Error of Mean 0.62

2. Primary Outcome: Personal Empowerment
Description: Personal psychological empowerment is measured via the Boston University Empowerment Scale (Rogers et al.,1997). This 28-item instrument designed to measure subjective feelings of empowerment via self-report in which respondents answer questions on a four-point scale ranging from Strongly Agree to Strongly Disagree. The minimum score is 28 and the maximum is 112, with higher scores indicating a better outcome.
Time Frame: Study entry (Pre-intervention/T1), 8-weeks later (Post-Intervention 1/T2), & 6-months after T2 (Post-Intervention 2/T3)
Population: The "Overall Number of Participants Analyzed" reflects the number of participants at Time 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BRIDGES Intervention | Comparison Wait-list Group
Number analyzed (Participants) | 212 | 216
score on a scale
  Baseline (Time 1) | 78.82 (9.29) | 78.58 (10.04)
  Post-intervention 1 (Time 2): number analyzed (Participants) | 171 | 172
  Post-intervention 1 (Time 2) | 82.31 (9.12) | 79.91 (9.88)
  Post-intervention 2 (Time 3): number analyzed (Participants) | 157 | 159
  Post-intervention 2 (Time 3) | 81.19 (9.21) | 79.57 (10.31)
Statistical Analysis 1: Comparison: BRIDGES Intervention vs Comparison Wait-list Group; We tested 3 moderating variables: BSI depressive symptom, anxiety, and general symptom distress. In these three models, we hypothesized that the intervention participants with high levels of each type of symptoms would experience greater gains in empowerment over time than participants with low levels of symptoms, as well as control participants with both high and low symptom level. This model includes depressive symptoms as the moderator (High depressive symptoms X time X study condition); Test type: Superiority; p = 0.01, Mixed Effects Random Regression; This analysis used Random Regression Modeling; this first model included depressive symptoms as moderator; MIXREG Estimate = 0.04, Standard Error of Mean .02
Statistical Analysis 2: Comparison: BRIDGES Intervention vs Comparison Wait-list Group; We tested 3 moderating variables: depressive symptom, anxiety, and general symptom distress. In these three models, we hypothesized that the intervention participants with high levels of each type of symptoms would experience greater gains in empowerment over time than participants with low levels of symptoms, as well as control participants with both high and low symptom level. This model includes anxiety as the moderator (high anxiety X time X study condition); Test type: Superiority; p = 0.01, Mixed Effects Random Regression; This analysis used Random Regression Modeling; this second model included anxiety symptoms as moderator; MIXREG Estimate = 0.04, Standard Error of Mean .02
Statistical Analysis 3: Comparison: BRIDGES Intervention vs Comparison Wait-list Group; We tested 3 moderating variables: BSI depressive symptom, anxiety, and general symptom distress. In these three models, we hypothesized that the intervention participants with high levels of each type of symptoms would experience greater gains in empowerment over time than participants with low levels of symptoms, as well as control participants with both high and low symptom level. This model includes general symptom distress as the moderator (high symptom distress X time X study condition); Test type: Superiority; p = .022, Mixed Effects Random Regression; This analysis used Random Regression Modeling; this third model included the general symptom distress as moderator; MIXREG Estimate = 0.03, Standard Error of Mean 0.01

3. Secondary Outcome: Hopefulness
Description: Hopefulness is measured by the State Hope Scale (Snyder et al., 1991). Hopefulness as a cross-situational long-term trait is assessed via patient self-report using a 12-item scale assessed on a 4-point Likert response scale with options ranging from "definitely false" to "definitely true" and summed to produce a total score and sub-scale scores. The minimum value for this scale is 12 and the maximum value is 48. Higher scores indicate a better income.
Time Frame: Study entry (Pre-intervention/T1), 8-weeks later (Post-Intervention 1/T2), & 6-months after T2 (Post-Intervention 2/T3)
Population: The "Overall Number of Participants Analyzed" reflects the number of participants at Time 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BRIDGES Intervention | Comparison Wait-list Group
Number analyzed (Participants) | 212 | 211
score on a scale
  Baseline | 22.64 (4.31) | 22.68 (4.77)
  Post-intervention 1 (Time 2): number analyzed (Participants) | 170 | 169
  Post-intervention 1 (Time 2) | 23.12 (3.73) | 22.77 (4.80)
  Post-intervention 2 (Time 3): number analyzed (Participants) | 155 | 159
  Post-intervention 2 (Time 3) | 23.24 (3.92) | 22.66 (4.73)
Statistical Analysis 1: Comparison: BRIDGES Intervention vs Comparison Wait-list Group; This mixed effects random regression analysis tested whether intervention participants would report larger increases than controls in Hopefulness that would be maintained longitudinally; Test type: Superiority; p < .01, Mixed Effects Random Regression; MIXREG Estimate = 0.33, Standard Error of Mean .012

4. Secondary Outcome: Patient Self-advocacy
Description: The ability to advocate for oneself with medical care providers is assessed via self-report using The Patient Self-Advocacy Scale (Brashers et al., 1999), an 18-item scale with a 5-point Likert response set ranging from "strongly disagree" to "strongly agree." Dimensions include in patient knowledge, assertiveness, and potential for mindful non-adherence to treatment. Scoring involves computing the mean scale score, so therefore values range from a minimum of 1 to a maximum of 5, with higher scores indicating a better outcome. Reported below are findings for the assertiveness sub-scale.
Time Frame: Study entry (Pre-intervention/T1), 8-weeks later (Post-Intervention 1/T2), & 6-months after T2 (Post-Intervention 2/T3)
Population: The Overall Number of Participants Analyzed reflects the number of participants at Time 1
Measure: Mean (Standard Deviation); unit: average score on a scale
Arm/Group | BRIDGES Intervention | Comparison Wait-list Group
Number analyzed (Participants) | 212 | 216
average score on a scale
  Baseline | 3.68 (0.71) | 3.72 (0.71)
  Post-intervention 1 (Time 2): number analyzed (Participants) | 171 | 171
  Post-intervention 1 (Time 2) | 3.82 (0.72) | 3.73 (0.76)
  Post-intervention 2 (Time 3): number analyzed (Participants) | 157 | 161
  Post-intervention 2 (Time 3) | 3.82 (0.73) | 3.79 (0.75)
Statistical Analysis 1: Comparison: BRIDGES Intervention vs Comparison Wait-list Group; This analysis Mixed Effects Random Regression Modeling to test whether self-advocacy scores changed overtime by study condition status. Reported below are findings for the self-advocacy assertiveness sub scale; Test type: Superiority; p < 0.01, Mixed Effects Random Regression; MIXREG Estimate = 0.12, Standard Error of Mean 0.04

5. Secondary Outcome: Coping Style
Description: Coping is measured via patient self-report using The Brief COPE Inventory (Carver, 1997), a 28-item instrument with 4-point Likert responses ranging from 1-"I haven't been doing this at all" to 4-"I have been doing this a lot." This measure includes two subscales that assess participants' adaptive coping skills (e.g., planning and using emotional support to deal with problems) and maladaptive coping skills (e.g., self-blame and denial). Scoring involves computing the means for each subscale, with a minimum value of 1 and a maximum value of 4. Higher adaptive coping scores indicate a greater use of positive coping styles; higher maladaptive coping scores indicate a greater use of negative coping styles (in other words, lower maladative coping scores indicate a better outcome).
Time Frame: Study entry (Pre-intervention/T1), 8-weeks later (Post-Intervention 1/T2), & 6-months after T2 (Post-Intervention 2/T3)
Population: The "Overall Number of Participants Analyzed" reflects the number of participants at Time 1. Results are provided for the Maladaptive Coping Subcale.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BRIDGES Intervention | Comparison Wait-list Group
Number analyzed (Participants) | 212 | 216
units on a scale
  Baseline (Time 1) | 2.14 (0.53) | 2.14 (0.54)
  Post-intervention 1 (Time 2): number analyzed (Participants) | 171 | 171
  Post-intervention 1 (Time 2) | 2.01 (0.51) | 2.13 (0.53)
  Post-intervention 2 (Time 3): number analyzed (Participants) | 157 | 161
  Post-intervention 2 (Time 3) | 2.04 (0.48) | 2.06 (0.52)
Statistical Analysis 1: Comparison: BRIDGES Intervention vs Comparison Wait-list Group; Test type: Superiority; p = 0.017, Mixed Effects Random Regression; MIXREG Estimate = 0.042, Standard Error of Mean .018

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a 2 year period.
Description: Adverse events in our behavioral health research study are indicated when participants report recent feelings of self-harm or harm to others either during the research interview assessments or at the time of an intervention.
Arm/Group | BRIDGES Intervention | Comparison Wait-list Group
All-Cause Mortality (participants affected / at risk) | 0/212 | 0/216
Serious Adverse Events (participants affected / at risk) | 0/212 | 0/216
Other Adverse Events (participants affected / at risk) | 1/212 | 2/216
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BRIDGES Intervention (N=212) | Comparison Wait-list Group (N=216)
Other Adverse Event (Psychiatric disorders) | 0 (0) | 1 (1) — 1 participant became upset and threatened self-harm because his money order received for completing his Time 2 interview was not able to be cashed at the currency exchange.The study's crisis protocol was activated and issue resolved.
Other Adverse Event (Psychiatric disorders) | 1 (1) | 0 (0) — At baseline interview, when asked questions from the Brief Symptom Inventory, a participant reported thoughts of suicide in the past 7 days. This occurred prior to start of intervention. The study's crisis protocol was activated.
Other Adverse Event (Psychiatric disorders) | 0 (0) | 1 (1) — At baseline interview, participant reported thoughts of self-harm during past week when asked questions from the Brief Symptom Inventory. The subject stated that he shares his feelings with therapist. The study's crisis protocol was also activated.

LIMITATIONS AND CAVEATS:
Limitations include recruitment from a single state rather than a nationally representative population, and reliance on self-report rather than clinician/researcher ratings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No